CLINICAL TRIAL: NCT03774693
Title: Efficacy of Regional Block of the Nose in Achieving Hypotensive Anaesthesia in Septo-rhinoplasty Surgery
Brief Title: Regional Block of the Nose for Hypotensive Anaesthesia in Septo-rhinoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanan Mahmoud Farag Awad, Assisstant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU R66/2018
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Hypotensive Anesthesia
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS [General anesthesia] (Active Comparator): Patients will receive general anesthesia with Fentanyl boluses of 0.5 mcg.Kg-1 given to maintain MAP between 55-65 mmHg with a maximum dose of 3 mcg.Kg-1.
  Interventions: Other: General anesthesia with fentanyl boluses
- GR [General anesthesia + regional block] (Active Comparator): Patients will receive general anesthesia with Fentanyl boluses of 0.5 mcg.Kg-1 given to maintain MAP between 55-65 mmHg with a maximum dose of 3 mcg.Kg-1.
  Also patients will receive trans-oral bilateral sphenopalatine ganglion block and trans-oral bilateral infraorbital nerve block. Fentanyl boluses of 0.5 mcg.Kg-1 will be given when needed to maintain MAP between 55-65 mmHg with a maximum dose of 3 mcg.Kg-1.
  Interventions: Other: General anesthesia with fentanyl boluses; Procedure: Regional block

INTERVENTIONS:
Other: General anesthesia with fentanyl boluses — Patients will receive general anesthesia with Fentanyl boluses of 0.5 mcg.Kg-1 given to maintain MAP between 55-65 mmHg with a maximum dose of 3 mcg.Kg-1
Procedure: Regional block — Patients will receive trans-oral bilateral sphenopalatine ganglion block and trans-oral bilateral infraorbital nerve block.
  Arms: GR [General anesthesia + regional block]

SUMMARY:
Septorhinoplasty is a cosmetic surgery that many people are choosing to undergo. It can be done under general anesthesia, twilight anesthesia or regional anesthesia. Controlled hypotensive anesthesia is required to minimize bruising, swelling, and bleeding that reduces visibility in the operative field and hence satisfactory surgical outcome.

The goal of our study to prove that regional block of the nose provides efficient hypotensive anesthesia

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II
* Scheduled for elective septo-rhinoplasty surgery

Exclusion Criteria:

* Patients with hypertension or coronary artery disease,
* Patients with renal, hepatic or cerebral insufficiency,
* Patients with coagulopathy or receiving drugs influencing blood coagulation,
* Patients with known sensitivity to any of the study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Hypotensive anesthesia | Intraoperative
  Measurement of Mean arterial blood pressure
Requirements of Fentanyl | Intraoperative
  Assessment of intraoperative fentanyl doses of [Fentanyl boluses of 0.5 mcg.Kg-1 will be given to maintain mean arterial pressure (MAP) between 55-65 mmHg with a maximum dose of 3 mcg.Kg-1]

SECONDARY OUTCOMES:
Average category scale (ACS) | Intraoperative
  The surgeon will be asked, at the end of surgery, to assess bleeding in the surgical field using the average category scale 0-5 scale where [0=No bleeding and5=Severe bleeding]

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided